CLINICAL TRIAL: NCT04346979
Title: The Effect of Telerehabilitation Based Yoga and Mindfulness Home Program on Psychological Resilience, Body Awareness and Physical Activity in Postmenopausal Women Having Social Isolation
Brief Title: Telerehabilitation-based Yoga and Mindfulness Home Program in Postmenopausal Women Having Social Isolation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istinye University (Other)
Responsible Party: Principal Investigator, Yasemin Çırak, Physiotherapist, PhD, Associate Professor, Istinye University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0001
Record Dates: First submitted 2020-04-13; First posted 2020-04-15 (Actual); Last update posted 2022-09-16 (Actual); Status verified 2022-09

CONDITIONS: Telerehabilitation
Keywords: Postmenopausal; Yoga; Mindfulness; COVID-19; Social Isolation
MeSH Terms: conditions — COVID-19; Social Isolation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group (Experimental): Telerehabilitation based yoga and mindfulness training will be given to the study group.
  Interventions: Other: Telerehabilitation-Based
- Control Group (Experimental): Yoga and mindfulness training will be provided by sending a video recording to the control group.
  Interventions: Other: Video-Based

INTERVENTIONS:
Other: Telerehabilitation-Based — 25 volunteers postmenopausal women who are at home during the social isolation process due to the coronavirus outbreak will be included in this group. Online yoga and mindfulness protocol was created for individuals who will participate in the study. Each training protocol was planned as 30 minutes for 3 days a week for 6 weeks. It was planned to start the protocol with warm-up exercises and finish with cooling exercises. Respiratory exercise was added to the training protocol. Individuals were asked to participate in the study via telerehabilitation system and aimed to do their exercises with a physiotherapist.
  Arms: Study Group
Other: Video-Based — 25 volunteers postmenopausal women who are at home during the social isolation process due to the coronavirus outbreak will be included in this group. Online yoga and mindfulness protocol was created for individuals who will participate in the study. Each training protocol was planned as 30 minutes for 3 days a week for 6 weeks. It was planned to start the protocol with warm-up exercises and finish with cooling exercises. The respiratory exercise was added to the training protocol. Video recordings containing only yoga and mindfulness training were sent to individuals. The participants were supervised by the researcher.
  Arms: Control Group

SUMMARY:
In the postmenopausal period when the woman spent 1/3 of her life; Due to the lack of estrogen, some physical and psychological changes occur. These changes may cause some problems. For women who perceive menopause as the first step of old age, loss of physical strength, energy, attraction and fertility, menopause can also lead to anxiety. In addition to these, they are among the emotional changes in the menopausal period in symptoms such as hypersensitivity to events, fatigue, and insomnia. Sometimes it can even be seen in psychological disorders such as melancholy and depression. The new coronavirus pneumonia (COVID-19), which appeared in Wuhan in December 2019, started to appear in different countries soon after. All countries have taken measures to prevent the spread of this virus. To this end, Turkey remains at home on March 21, 2020, and has commissioned social isolation measures. Studies investigating the effects of social isolation show that psychological and physical problems occur in individuals. Studies have shown that yoga and mindfulness programs have an impact on people's anxiety, depression, and the ability to control themselves. The purpose of this study; To investigate the effectiveness of telerehabilitation based yoga and mindfulness programs on psychological resilience, physical awareness and physical activity in postmenopausal women in social isolation due to the COVID-19 outbreak. Using telerehabilitation-based home programs aims to use an innovative model.

ELIGIBILITY:
Inclusion Criteria:

* Being physically or perceptually competent to exercise,
* No spinal pathology or deformity,
* Volunteering to participate in the study,
* Not having menstruation for at least 12 months
* Hormonally, surgically induced or natural menopause-confirmed women

Exclusion Criteria:

* Those with serious heart disease (aortic stenosis, angina, hypertrophic cardiac myopathy, arrhythmia, pacemaker)
* Those with inflammatory or systemic disease malignancy
* Psychological dysfunction
* Those who use corticosteroids

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 50 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-11-01 (Actual)

PRIMARY OUTCOMES:
The Brief Resilience Scale | 2 week
  The scale was used to measure the psychological resilience of individuals and Smith et al. (2008) were developed by. It is a 5-point Likert type, 6-item self-reporting style measurement tool. After the items in the scale and reverse coded are translated, the high scores indicate high psychological soundness.
Nottingham Health Profile | 2 week
  Nottingham Health Profile was created in England in 1985 to evaluate the quality of life-related to health. The Nottingham Health Profile is a general quality of life questionnaire that assesses the level of individuals health problems and how they affect their daily life activities.
Mindful Attention Awareness Scale | 2 week
  Mindful Attention Awareness Scale developed by Brown and Ryan (2003) is a 15-item scale that measures the general tendency to be aware of and be mindful of instant experiences in daily life. It has a single factor structure and gives a single total score. High scores from the scale indicate that conscious awareness is high. It is a 6-point Likert type scale.
The Body Awareness Questionnaire | 2 week
  It is a questionnaire consisting of four subgroups (changes in body process, sleep-wake cycle, prediction at the onset of the disease, prediction of body responses) and a total of 18 expressions aimed at determining the normal or abnormal sensitivity level of the body composition. The participant is asked to score from one to seven figures for each statement. In the survey, the ratings are made as total points. A high score indicates that body sensitivity is better.
Richard-Campbell Sleep Questionnaire | 2 week
  It, developed by Richards in 1987, is a 6-item scale that evaluates the depth of night sleep, falling asleep, frequency of waking, awakening when awakened, the quality of sleep and the level of noise in the environment. Each item is evaluated on the chart between 0 and 100 with a visual analog scale technique. "0-25" score obtained from the scale indicates very poor sleep, and the "76-100" score indicates very good sleep. Scale total score is evaluated over 5 items, and item 6 evaluating the noise level in the environment is excluded from the total score assessment. As the score of the scale increases, the sleep quality of the patients also increases.
Lateral bridge test | 2 week
  The participant, who is on the non-dominant side, will be asked to create a support surface from the elbow with the lower arm, place the other hand on the waist, and build a bridge by lifting the hip and knee. The time that the balance is maintained will be recorded.
Functional reach test | 2 week
  It is applied functionally both for the balance of the individual and for measuring the amount of dynamic reach. The individual is asked to lie down as long as he/she can lie down without going over the heel and hip flexion.
Beck Depression Scale | 2 week
  It consists of 21 questions used to evaluate the emotional situation. Each question is graded between 0-3 and a high score indicates that depressive symptoms increase. 10-16 points indicate mild depressive symptoms, 17-29 points indicate moderate depressive symptoms and 30-63 points indicate severe depressive symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Istinye University, Istanbul, Turkey (Türkiye)